CLINICAL TRIAL: NCT02621125
Title: Fertilix Supplements and Assisted Reproductive Technology
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Reproductive Associates (Other)
Collaborators: CellOxess LLC (Industry)
Responsible Party: Principal Investigator, Peter McGovern, MD, Principal Investigator, University Reproductive Associates
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Fertilix
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Spermatozoa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fertilix (Experimental): Fertilix supplementation
  Interventions: Dietary Supplement: Fertilix
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Fertilix — daily supplementation
  Arms: Fertilix
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a double blind, randomized, placebo controlled clinical trial to test the efficacy of the antioxidant formulation Fertilix® in lowering the levels of damaged sperm DNA in men diagnosed with moderate to high Sperm Oxidative DNA Damage (SODD)

ELIGIBILITY:
Inclusion Criteria:

* Males with a sperm sample containing 8-OHdG levels > 15% and must be capable of producing an ejaculate containing >10million sperm upon study enrollment.
* Male is between 20-55 years of age seeking treatment for infertility with his partner at URA and who is a candidate for an IUI, IVF or IVF-ICSI (excluding donor egg) procedure.
* Female is between 20-42 years of age
* Female exhibits tubal patency on hydrosonogram or hysterosalpingogram (HSG)
* Female exhibits normal uterine cavity by hysteroscopy, hydrosonogram or hysterosalpingogram (HSG).

Exclusion Criteria

* Subjects with initial semen analysis of an ejaculate containing < 10 million sperm.
* Men who have been taking nutraceuticals, vitamins or other compounds known to have antioxidant activities within4 weeks of the study. No other supplements may be taken with Fertilix.
* Men who have hypersensitivity or an allergy to any of the ingredients in Fertilix®.
* Men who have been treated with a chemotherapeutic agent known to cause sterility, such as cyclophosphamide.
* Men who have taking anabolic steroids or testosterone replacement within 4 months of the study.
* Men currently being treated with a Ca++ channel blocker or other medical treatment known to adversely affect sperm production or function.
* Men with HIV, hepatitis B and C.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Reduction in sperm DNA damage | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Reproductive Associates, Hasbrouck Heights, New Jersey, United States